CLINICAL TRIAL: NCT06996808
Title: Intrauterine Balloon (Bakri©) Versus Uterine Tamponade With Chitosan Gauze (Celox PPH©) in the Management of Postpartum Hemorrhage Refractory to Medical Treatment: A Multicenter Randomized Controlled Trial
Brief Title: Intrauterine Balloon (Bakri©) Versus Uterine Tamponade With Chitosan Gauze (Celox PPH©) in the Management of Postpartum Hemorrhage Refractory to Medical Treatmen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Rizzo, Full Professor Obstetrics and Gynecology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 400/8.04.2025 4a4
Record Dates: First submitted 2025-05-12; First posted 2025-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : Bakri Balloon (Active Comparator): Bakri Balloon Standard insertion and inflation as per hospital protocol following delivery.
  Interventions: Device: Bakri Baloon
- : Celox Gauze (Experimental): Celox gauze will be placed intrauterine according to manufacturer instructions, post-vaginal or cesarean delivery. Duration and removal will follow standardized clinical guidelines.
  Interventions: Device: Celox gauze

INTERVENTIONS:
Device: Bakri Baloon — Bakri Balloon Standard insertion and inflation as per hospital protocol following delivery.
  Arms: : Bakri Balloon
Device: Celox gauze — Celox gauze will be placed intrauterine according to manufacturer instructions, post-vaginal or cesarean delivery. Duration and removal will follow standardized clinical guidelines
  Arms: : Celox Gauze

SUMMARY:
Postpartum hemorrhage (PPH) remains one of the leading causes of maternal morbidity and mortality worldwide, particularly in low- and middle-income countries. It is defined as blood loss of more than 500 mL after vaginal delivery or more than 1000 mL after cesarean section, but severe PPH is typically identified when blood loss exceeds 1000 mL regardless of delivery mode. The initial management of PPH includes the administration of uterotonics such as oxytocin, methylergometrine, and tranexamic acid. However, a subset of patients remains unresponsive to medical therapy, necessitating second-line interventions to avoid escalation to invasive procedures such as uterine artery embolization or peripartum hysterectomy.

An intrauterine balloon tamponade device (Bakri©), is commonly used as a mechanical method to control uterine bleeding by exerting direct pressure on the uterine walls. Its use has been widely adopted and incorporated into international guidelines due to its relative ease of use and safety profile. Despite its effectiveness, the failure rate of Bakri balloon placement can range from 20% to 40%, especially in cases of coagulopathy or diffuse atony.

Gauzes with a chitosan-based hemostatic dressing (Celox PPH ©) , has been extensively used in trauma settings and is increasingly being explored for surgical and obstetric applications. Its mechanism involves promoting clot formation independent of the clotting cascade, making it potentially beneficial in patients with coagulopathies. Preliminary data and case reports suggest that Celox PPH© may be effective in controlling intrauterine bleeding when used as a packing material after vaginal or cesarean delivery, but no high-quality randomized controlled trial has yet compared it directly with standard interventions.

Given the clinical need for alternative second-line treatments for PPH unresponsive to medical therapy, this study proposes a head-to-head comparison of the Bakri balloon and Celox gauze. The findings will help inform evidence-based guidelines and may offer new strategies to reduce maternal transfusion requirements, prevent hysterectomy, and shorten hospital stays in patients experiencing severe PPH.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following criteria to be eligible for inclusion:

* Women aged 18 years or older who have delivered either vaginally or via cesarean section.
* Diagnosis of postpartum hemorrhage, defined as an estimated blood loss (EBL) greater than 1000 mL within the first 24 hours postpartum.
* Refractory to first-line medical therapy, specifically high-dose oxytocin (≥40 IU total administered intravenously or intramuscularly), a full dose of methylergometrine (0.2 mg IM or IV), and administration of tranexamic acid (1 g IV).
* Hemodynamically stable at the time of enrollment, allowing time for the application of a mechanical or topical intervention.

Exclusion Criteria: Patients will be excluded if they meet any of the following conditions:

* Clinical or radiological suspicion of placenta accreta spectrum (PAS), including placenta increta or percreta, which may necessitate immediate surgical management.
* Known pre-existing or newly diagnosed coagulopathy, including but not limited to thrombocytopenia (<50,000/μL), von Willebrand disease, hemophilia, or disseminated intravascular coagulation (DIC), which may compromise the safety or efficacy of the interventions.
* Hemodynamic instability defined by persistent hypotension (systolic BP <90 mmHg or MAP <65 mmHg) despite resuscitation, or active decision to proceed to surgical intervention (e.g., laparotomy, uterine artery embolization, or hysterectomy) without delay.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin levels | From enrollment to 24 hours after delivery
  Materal hemoglobin levels will be assessd at diagnosis of Post partum hemorrage, 24 after delievry and at the discharge
Needs of blood transfusion | From enrollment to 24 hours after delivery

SECONDARY OUTCOMES:
Hysterectomy | From enrollment to one week after delivery
  Need of performing hysterectomy
Lenght of hospital stay | From delivery up to 6 weeks postpartum
ICU admission | From enrollment up to 6 weeks postpartum
Need for surgical intervention | From enrollment to the firstday after delivery and at one week
  needs of other surgical procedures (i.e, suture of uterine lacerations, uterine hemostatic suture(ì)

IPD SHARING:
Plan to Share IPD: Undecided